CLINICAL TRIAL: NCT04143789
Title: A Phase 1/2 Dose Escalation Study of AP-002 In Patients With Advanced or Recurrent Solid Tumors
Brief Title: Evaluation of AP-002 in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Altum Pharmaceuticals INC (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALT-002-SRE-01
Record Dates: First submitted 2019-10-04; First posted 2019-10-29 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Review of safety and pharmacokinetic (PK) parameters by the Clinical Trial Review Committee (CTRC) at the completion of each dose level in the Phase 1 will determine if escalation to the next dose level may occur.
  Anticipated Dose Levels in the Phase 1 Portion of the Study Cohort Anticipated Dose Anticipated Sample Size Level 1 8 mg QD PO × 14 days* (1 patient) Level 2 16 mg QD PO × 14 day* (1 patient) Level 3 32 mg QD PO × 14 days* (1 patient) Level 4 64 mg QD PO × 14 days* (1 patient) Level 5 84 mg QD PO × 14 days* (3 patients) Level 6 108 mg QD PO × 14 days* (3 patients) Level 7 140 mg QD PO × 14 days* (3 patients) Level 8 180 mg QD PO × 14 days* (3 patients)
  * Note: 21-day schedule with 2 weeks on, one week off. The actual sample size will be guided by the CRM; sample size may be larger for dose levels that require expansion. Interim meetings may occur when relevant new data becomes available between scheduled CTRC meetings
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tablets to be taken orally daily for 14 of 21 day cycle (Experimental): AP-002 (4 mg and 20 mg tablets) to be taken orally daily for 14 days
  Interventions: Drug: AP-002

INTERVENTIONS:
Drug: AP-002 — Dose escalation
  Other Names: no other names

SUMMARY:
The purpose of this trial is to define an effective and safe dose of AP-002 in advanced or recurrent solid tumors for which there are no standard therapies to use in subsequent studies in advanced or recurrent breast, non-small cell lung cancer (NSCLC) or prostate cancers.

DETAILED DESCRIPTION:
The Phase 1 portion of this study will determine the Pharmacodynamically Active Dose (PAD) of AP-002 in humans, defined as the dose at which the plasma concentration of AP-002, as measured by Ga, is 300-500 ng/mL and which is at or below the Maximum Tolerated Dose (MTD), to use in the clinical setting of advanced or recurrent solid tumors. This will be followed by a Phase 2 expanded cohort treated at the PAD, to estimate the efficacy of AP-002 in patients with advanced or recurrent breast cancer, NSCLC and prostate cancer.

Patients will receive AP-002 orally, once daily for 14 days of a 21 day cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1: Patients with advanced or recurrent solid tumors with target (± non-target) or with only non-target disease, for which there is no standard therapy available Phase 2: Patients with advanced or recurrent breast cancer, NSCLC, or prostate cancer with target (± non-target) or with only non-target disease for which there is no standard therapy available
2. Patients with bone metastases but without target disease are eligible
3. Patients with bone metastases must have at least one bone lesion that has not received radiation therapy within 6 weeks prior to Cycle 1 Day 1
4. Patients must discontinue bisphosphonate and/or denosumab treatment.
5. Age ≥ 18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
7. O2 saturation ≥ 92% on room air per pulse oximetry
8. Exhaled nitrous oxide ≤ 50 parts per billion (ppb)
9. Adequate hematologic, hepatic and renal function defined as:

   1. Hemoglobin ≥ 9 g/dL
   2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
   3. Platelet count ≥ 75 × 109/L
   4. Total bilirubin ≤ 2 × upper limit of normal (ULN). Patients with an established diagnosis of Gilberts syndrome with an unconjugated bilirubin ≤ 2 mg/dL and conjugated bilirubin within normal limits (WNL) are eligible.
   5. Serum electrolytes WNL
   6. Transaminases ≤ 3 × ULN
   7. Prothrombin time (PT)/international normalized ratio (INR), thromboplastin time (PTT), or activated PTT (aPTT) ≤ 1.5 × ULN. For patients on therapeutic coumadin, PT (INR) ≤ 2.5 × ULN is acceptable; for patients on therapeutic heparin, PTT (or aPTT) ≤ 2.5 × ULN
   8. Corrected creatinine clearance ≥ 40 mL/minute, based on the Cockcroft-Gault equation
10. Patient must have discontinued prior antineoplastic therapy at least 21 days prior to Cycle 1 Day 1 and have recovered or stabilized from any prior AEs related to the prior therapy
11. Provision of signed and dated informed consent form
12. Serum 25-hydroxyvitamin D ≥ 30 ng/mL by investigative site laboratory at screening

Exclusion Criteria:

1. Evidence of benign primary hyperparathyroidism, hyperthyroidism, adrenal insufficiency, vitamin D intoxication, mild alkali syndrome, sarcoidosis or other granulomatous disease
2. Treatment with calcitonin, mithramycin or cinacalcet within 7 days prior to the date of the screening
3. Receiving dialysis for renal failure
4. Patients with a known history of clinically significant active infection, including human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
5. Patients with active central nervous system (CNS) metastases are not eligible, but patients with treated, stable CNS metastases are allowed
6. Patients with QT interval of ≥ 480 msec on ECG
7. Patients with Paget's disease of bone
8. Patients of childbearing potential unwilling to abstain from sexual intercourse, or employ effective barrier methods of contraception during participation in this trial
9. Pregnancy or lactation. A negative pregnancy test will be required for women of childbearing potential prior to study enrollment and will be repeated throughout the study. Women of childbearing potential will be defined as women who have not had natural or pharmacologic menopause, nor surgical sterilization.
10. Patients unwilling or unable to take oral medication, requiring a nasogastric or gastrostomy tube, or unwilling to adhere to the treatment regimen and fasting requirements
11. Patients unwilling to comply with all study procedures or who are unavailable for the duration of the study
12. Known allergies to any components of the AP-002 Drug Product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment | Through study completion/ up to 18 months
  Number of participants with treatment-related adverse events (safety and tolerability) as assessed by CTCAE v4.0
Dose Assessment | Up to 6 months
  Define the recommended phase 2 dose

SECONDARY OUTCOMES:
Efficacy Assessment | Through study completion/ up to 18 months
  Estimation of anti-tumor activity per RESIST v1.1
Efficacy Assessment | Through study completion/ up to 18 months
  For patients with bone metastases, the time to new bone metastasis, progression of bone metastases, or other skeletal related events
Pharmacokinetic Assessment | Through study completion/ up to 18 months
  Estimation of pharmacokinetic profile by evaluating maximum plasma concentration [Cmax]

CONTACTS AND LOCATIONS:
Overall Officials: Angela Ogden, MD, Study Chair — Altum Pharmaceuticals
Locations (3):
- United States (3):
  - Research Institution, Chicago, Illinois
  - Research Site, St Louis, Missouri
  - Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Diaries will be left at site and used as source documents